CLINICAL TRIAL: NCT03051802
Title: Feasibility Study of Navigated Endoscopy for the Placement of High Dose Rate Brachytherapy Applicators in the Esophagus and Lung
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-5056
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Esophagus Cancer; Lung Cancer
Keywords: Endoscopy; HDR Brachytherapy; navigation
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Navigated Endoscopy — Navigated endoscopy used to guide the placement of HDR applicators in the esophagus or lung as a replacement to current standard of practice using fluoroscopic imaging.

SUMMARY:
The scope of this clinical trial is to assess the clinical feasibility of this procedure, optimize the protocol and perform an initial comparison of the positional accuracy of navigated endoscopy and applicator insertion versus the standard of care 2D fluoroscopy protocol.

DETAILED DESCRIPTION:
High dose rate brachytherapy is used in a limited number of esophagus and lung patients, often in combination with external beam radiation therapy. The procedure uses an applicator inserted into the lumen with the applicator connected to an automated "afterloader", a device with a radioactive brachytherapy source attached to a thick guide wire that positions the source within the applicator at set positions and times based on a treatment plan. Identification of the ideal applicator position is determined by white light endoscopy. With the endoscope in the lumen, fluoroscopic imaging can visualize the endoscope position. Temporary radio-opaque skin markers are placed on the patient's anterior surface under fluoroscopy imaging so that they align with the endoscope tip. The proximal and the distal ends of the target volume are marked in this manner by the surgeon stopping the endoscope at these positions. The endoscope is removed and the applicator inserted, with the positions of the applicator and "dummy" seeds (i.e. non-radioactive seeds used only for positioning purposes) aligned under fluoroscopy to match the skin markers. The procedure has 2 disadvantages: i. There is extra radiation dose to the clinical staff due to the fluoroscopy used to identify the source position.

ii. Visualization is only in 2D, which is inaccurate since it does not account for separations in the vertical direction and the angle of projection between the applicator and the so patient surface. Furthermore, any movement of the fluoroscopy device during the insertion leads to errors in visualization.

Medical applications of navigated endoscopy continue to grow, especially when used in combination with volumetricimaging for image-guided procedures. This feasibility study is aimed to use navigation endoscopy technology to overcome the disadvantages of the current practice and improve the overall process.

In the proposed protocol, applicator insertion, tracking and recording of the endoscope and applicator positions would enable placement of the applicator using 3D information, with greater accuracy and without extra radiation dose to the clinical staff. The tracking technology would be used to replace the use of radio-opaque skin markers; rather than placing these markers on the patient's skin, the location of the target volume boundaries would be noted by the tracker position within the endoscope. Applicator insertion would also be tracked, with the applicator positioning based on the location of the applicator relative to the previously recorded endoscope positions, including the locations of the distal and proximal ends of the target volume.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary or metastatic cancer including endoluminal disease of either the lung or the esophagus
* Intention to treat using high dose rate brachytherapy as part of standard radiotherapy.
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Contraindications to standard radiation therapy including pregnancy, lactation, connective tissue disorders, serious co-morbid illness
* Concurrent illness or condition that precludes subject from undergoing endoscopy
* Patient is unable to tolerate an hour and a half long procedure. Standard of care practice is no more than 1 hour. However, with the additional tracking component, the procedure could be at most 1.5 hours long.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
proportion of navigated endoscopy procedures that were successfully completed | 18 months
  To assess clinical feasibility of inserting intraluminal (esophagus or lung) HDR applicators using navigation technologies for tracking endoscope and applicator insertion.
  This study is designed to assess the workflow when using the EM tracking technology and the accuracy of the procedure will be measured by comparison with current standard of care.
Positional accuracy | day 1
  To compare the positional accuracy of the navigation procedure versus the current standard of care using 2D fluoroscopy using analysis of tracking data. All tracking data will be recorded for post-procedure analysis and comparison with the fluoroscopic imaging performed during current standard of care
Optimize the clinical protocol using this technology | 6 months
  The procedure will be assessed in detail (based on time and workflow) after three patients. Participants in the review of the procedure will include surgeon, radiation oncologist, brachy-therapists and physicists. Workflow improvements will be implemented at this time.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No